CLINICAL TRIAL: NCT01322971
Title: Pregnancy Outcomes Following Preconception Treatment of Asymptomatic Bacterial Vaginosis in an Infertility Population: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial.
Brief Title: Efficacy Study of Preconception Treatment of an Asymptomatic Bacterial Infection in an Infertility Population
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Disease prevalence lower than expected in population.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ruth Bunker Lathi, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-03212011-7604; IRB Protocol Number 20103 (Other: Stanford IRB)
Record Dates: First submitted 2011-03-23; First posted 2011-03-25 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Vaginosis, Bacterial; Infertility; Miscarriage
Keywords: Bacterial Vaginosis; Infertility; Miscarriage; Metronidazole
MeSH Terms: conditions — Vaginosis, Bacterial; Infertility; Abortion, Spontaneous | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metronidazole (Active Comparator): Patients randomized to the metronidazole arm will receive metronidazole 500mg orally twice daily for seven days.
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Patients randomized to the placebo arm will receive placebo orally twice daily for seven days(control arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — Metronidazole 500mg orally twice daily for seven days
  Arms: Metronidazole
Drug: Placebo — Placebo will be administered orally twice daily for seven days
  Arms: Placebo

SUMMARY:
Bacterial vaginosis (BV) is a common vaginal infection characterized by a pathologic shift in the normal vaginal flora. BV has been associated with a number of poor reproductive outcomes, including infertility, preterm labor and premature rupture of membranes. If BV does disrupt normal embryologic development, then the treatment of BV prior to conception may improve implantation rates and other pregnancy outcomes in the infertile population.

This is a prospective, randomized, double-blind, placebo-controlled trial in which infertile women undergoing intrauterine insemination or embryo transfer are screened for BV prior to treatment. Those patients who screen positive for BV will then be randomized into the treatment arm(metronidazole 500mg by mouth twice daily for 7 days) or the control arm (placebo by mouth twice daily for 7 days). The primary outcome, positive pregnancy test rate (i.e. biochemical pregnancy rate), will then be assessed. Secondary outcomes, such as clinical pregnancy rate, miscarriage rate, and live birth rate will also be examined.

DETAILED DESCRIPTION:
The purpose of this study is to determine if preconception treatment of asymptomatic bacterial vaginosis improves pregnancy outcomes (i.e. biochemical pregnancy rate). Study protocol as follows:

1. Patients will be notified of study via face-to-face contact at the initial clinic visit (baseline ultrasound visit, menstrual cycle day 2-5), by physician referral or the Stanford website. Patients expressing interest will be screened in person to confirm that they meet all enrollment criteria. The participant will be asked to sign informed consent documents and a brief intake questionnaire with then be administered.
2. Enrolled patients will then be screened for bacterial vaginosis at their next visit (typically on menstrual cycle day 12), prior to transvaginal ultrasound. The screening will require that a speculum be inserted into the vagina and a vaginal smear be collected with a swab from the posterior fornix. A microscopic slide will be prepared by rolling the swab on the surface of a glass slide. The diagnosis of bacterial vaginosis will be established clinically using the Amsel criteria to confirm 3 of the following 4 signs: clue cells; vaginal pH ≥4.5; fishy odor before or after the addition of 10% potassium hydroxide solution to a wet-mount side; and a homogeneous, off-white, discharge. For validation of clinical diagnosis, 100% of screen positive slides, and 10% of screen negative slides, will be sent for to the Department of Pathology for Gram staining.
3. The patients with a positive screen for bacterial vaginosis will then be randomized to receive metronidazole 500mg orally twice daily for seven days (treatment arm) or placebo orally twice daily for seven days(control arm). Randomization will be performed using a computer-generated code. Those patients whose screen is negative will also be followed for outcomes, but no randomization will be performed.
4. All randomized patients will continue with routine monitoring and insemination as planned by their treating physician.
5. If pregnancy is confirmed at least 12 weeks after intrauterine insemination by ultrasound evidence of a fetus with heartbeat, information will then be collected regarding the pregnancy and its outcome.
6. Primary and secondary outcomes will be followed for 2 years after date of enrollment for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Women who are actively trying to conceive via intrauterine insemination or in vitro fertilization

Exclusion Criteria:

* Current use of an oral or vaginal antibiotic.
* History of allergy or adverse reaction to metronidazole.
* Prior enrollment in study (patients returning for repeat cycle may not be re-enrolled).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Bunker Lathi, Principal Investigator — Stanford University
Locations (1):
- Ruth Lathi, Stanford, California, United States

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin. Assessment of risk factors for preterm birth. Clinical management guidelines for obstetrician-gynecologists. Number 31, October 2001. (Replaces Technical Bulletin number 206, June 1995; Committee Opinion number 172, May 1996; Committee Opinion number 187, September 1997; Committee Opinion number 198, February 1998; and Committee Opinion number 251, January 2001). Obstet Gynecol. 2001 Oct;98(4):709-16. PMID 11592272
- [Background] Carey JC, Klebanoff MA, Hauth JC, Hillier SL, Thom EA, Ernest JM, Heine RP, Nugent RP, Fischer ML, Leveno KJ, Wapner R, Varner M. Metronidazole to prevent preterm delivery in pregnant women with asymptomatic bacterial vaginosis. National Institute of Child Health and Human Development Network of Maternal-Fetal Medicine Units. N Engl J Med. 2000 Feb 24;342(8):534-40. doi: 10.1056/NEJM200002243420802. PMID 10684911
- [Background] Donders GG, Van Bulck B, Caudron J, Londers L, Vereecken A, Spitz B. Relationship of bacterial vaginosis and mycoplasmas to the risk of spontaneous abortion. Am J Obstet Gynecol. 2000 Aug;183(2):431-7. doi: 10.1067/mob.2000.105738. PMID 10942482
- [Background] Hay PE, Lamont RF, Taylor-Robinson D, Morgan DJ, Ison C, Pearson J. Abnormal bacterial colonisation of the genital tract and subsequent preterm delivery and late miscarriage. BMJ. 1994 Jan 29;308(6924):295-8. doi: 10.1136/bmj.308.6924.295. PMID 8124116
- [Background] Hay PE. Bacterial vaginosis and miscarriage. Curr Opin Infect Dis. 2004 Feb;17(1):41-4. doi: 10.1097/00001432-200402000-00008. PMID 15090889
- [Background] Hillier SL, Nugent RP, Eschenbach DA, Krohn MA, Gibbs RS, Martin DH, Cotch MF, Edelman R, Pastorek JG 2nd, Rao AV, et al. Association between bacterial vaginosis and preterm delivery of a low-birth-weight infant. The Vaginal Infections and Prematurity Study Group. N Engl J Med. 1995 Dec 28;333(26):1737-42. doi: 10.1056/NEJM199512283332604. PMID 7491137
- [Background] Korn AP, Bolan G, Padian N, Ohm-Smith M, Schachter J, Landers DV. Plasma cell endometritis in women with symptomatic bacterial vaginosis. Obstet Gynecol. 1995 Mar;85(3):387-90. doi: 10.1016/0029-7844(94)00400-8. PMID 7862377
- [Background] Liversedge NH, Turner A, Horner PJ, Keay SD, Jenkins JM, Hull MG. The influence of bacterial vaginosis on in-vitro fertilization and embryo implantation during assisted reproduction treatment. Hum Reprod. 1999 Sep;14(9):2411-5. doi: 10.1093/humrep/14.9.2411. PMID 10469722
- [Background] McDonald HM, Brocklehurst P, Gordon A. Antibiotics for treating bacterial vaginosis in pregnancy. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD000262. doi: 10.1002/14651858.CD000262.pub3. PMID 17253447
- [Background] Nelson DB, Bellamy S, Nachamkin I, Ness RB, Macones GA, Allen-Taylor L. First trimester bacterial vaginosis, individual microorganism levels, and risk of second trimester pregnancy loss among urban women. Fertil Steril. 2007 Nov;88(5):1396-403. doi: 10.1016/j.fertnstert.2007.01.035. Epub 2007 Apr 16. PMID 17434499
- [Background] Platz-Christensen JJ, Brandberg A, Wiqvist N. Increased prostaglandin concentrations in the cervical mucus of pregnant women with bacterial vaginosis. Prostaglandins. 1992 Feb;43(2):133-4. doi: 10.1016/0090-6980(92)90082-5. PMID 1542740
- [Background] Platz-Christensen JJ, Mattsby-Baltzer I, Thomsen P, Wiqvist N. Endotoxin and interleukin-1 alpha in the cervical mucus and vaginal fluid of pregnant women with bacterial vaginosis. Am J Obstet Gynecol. 1993 Nov;169(5):1161-6. doi: 10.1016/0002-9378(93)90274-m. PMID 8238178
- [Background] Wilson JD, Ralph SG, Rutherford AJ. Rates of bacterial vaginosis in women undergoing in vitro fertilisation for different types of infertility. BJOG. 2002 Jun;109(6):714-7. doi: 10.1111/j.1471-0528.2002.01297.x. PMID 12118653

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 151 participants were screened ; 2 were randomized
Period: Overall Study
Arm/Group | Metronidazole | Placebo
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 37 (0) | 37 (0) | 37 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Pregnancy Rate (Positive Pregnancy Test)
Description: Biochemical pregnancy rate was defined as number of participants who had a positive pregnancy test
Time Frame: up to 2 years
Population: No data were collected for this outcome
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pregnancy Rate (Pregnancy Visible on Ultrasound)
Time Frame: up to 2 years
Population: No data were collected for this outcome
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Miscarriage Rate (Loss of a Clinically Recognized Pregnancy)
Time Frame: up to 2 years
Population: No data were collected for this outcome
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Infectious Morbidity (i.e. Chorioamnionitis, Neonatal Sepsis)
Time Frame: up to 2 years
Population: No data were collected for this outcome
Arm/Group | Metronidazole | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: All participants withdrew prior to entering any protocol specified adverse event collection period.
Arm/Group | Metronidazole | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
151 screened 2 were randomized both refused to take medication not knowing if it were placebo or drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No